CLINICAL TRIAL: NCT07028736
Title: Assessment of Dry Eye Disease and Retinal Nerve Fiber Layer Thickness in Chronic Smokers
Brief Title: Dry Eye Disease and Retinal Nerve Fiber Layer Thickness in Chronic Smokers
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Merna Tharwat Wanees Nakhla, Resident of Ophthalmology, Faculty of Medicine, Cairo University, Cairo, Egypt., Cairo University
Other Study IDs: MS-250-2023
Record Dates: First submitted 2025-06-03; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Dry Eye Disease; Retinal Nerve Fiber Layer; Chronic Smoking
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Non-smokers.
  Interventions: Other: Dry eye assessment
- Group B: Chronic smokers (≥1 pack/day for ≥10 years).
  Interventions: Other: Dry eye assessment

INTERVENTIONS:
Other: Dry eye assessment — Dry eye assessment was performed using the Mediworks Dry Eye Diagnostic System.

SUMMARY:
This study aimed to examine the impact of long-term smoking on dry eye parameters and retinal nerve fiber layer thickness in individuals who are chronic smokers.

DETAILED DESCRIPTION:
Dry eye disease (DED) is a multifaceted disorder of the ocular surface characterized by instability of the tear film, which subsequently leads to symptoms such as ocular discomfort, visual disturbances, and potential damage to the surface of the eye.

Cigarette smoking has been recognized as a possible contributing factor to the development of DED, with various reports suggesting that it may alter tear film composition and stability, leading to ocular surface damage.

Chronic smoking can lead to oxidative stress, vascular dysfunction, and inflammation, which may contribute to retinal nerve fiber layer (RNFL) thinning and optic nerve damage.

ELIGIBILITY:
Inclusion Criteria:

* Age from 30 to 60 years.
* Both sexes.
* Chronic smokers.

Exclusion Criteria:

* History of ocular surface diseases affecting tear production or secretion (such as Sjogren's syndrome or Stevens-Johnson disease).
* Conjunctivitis.
* Blepharitis.
* Chronic contact lens use or gross lid abnormalities.
* Preexisting glaucoma.
* Retinal diseases.
* Optic nerve pathology.
* Ocular trauma.
* Chemical burns.
* Recent eye surgery (within three months).
* Trachoma-related complications

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This observational case-control study was conducted on a total of 100 eyes from 50 patients.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Non-invasive tear film breakup time | During examination (Baseline)
  Non-invasive tear film breakup time (NIBUT) was automatically analyzed using artificial intelligence, with results classified as Grade 0 (normal, first rupture time >10s), Grade 1 (warning, 6- 9s), or Grade 2 (dry eye, ≤5s)

SECONDARY OUTCOMES:
Tear meniscus height | During examination (Baseline)
  Tear meniscus height (TMH) values above 0.2mm were considered healthy, while lipid layer thickness was graded from 1 (<30nm) to 4 (>80nm).
Lipid layer thickness | During examination (Baseline)
  Lipid layer thickness was graded from 1 (<30nm) to 4 (>80nm).
Ocular Surface Disease Index (OSDI) score | During examination (Baseline)
  The ocular surface disease index (OSDI) score was categorized as normal (≤12), mild (13-22), moderate (23-32), or severe (≥33).
Retinal nerve fiber layer thickness | During examination (Baseline)
  Retinal nerve fiber layer (RNFL) thickness was measured using Fourier-domain OCT Optovue RTVue (Optovue Inc., Fremont, CA, USA).
Correlations between dry eye parameters and Ocular Surface Disease Index (OSDI) score | During examination (Baseline)
  Correlations between dry eye parameters and Ocular Surface Disease Index (OSDI) score was assessed.
Correlations between dry eye parameters and retinal nerve fiber layer (RNFL) thickness in both groups | During examination (Baseline)
  Correlations between dry eye parameters and retinal nerve fiber layer (RNFL) thickness in both groups was assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.